CLINICAL TRIAL: NCT04846660
Title: Examining the Impact of Production Pressure in the Regional Anesthesia Block Room on Patient Safety, a Randomized Single Blind Study in a High Fidelity Simulation Environment
Brief Title: Impact of Production Pressure in the Block Room on Patient Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Université de Montréal (Other); Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Marie-Eve Belanger, Associate Professor, MD, FRCPC, PGdip(ed), Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-2533
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Patient Safety; Anesthesia
Keywords: Production pressure; Time pressure
MeSH Terms: conditions — Time Pressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blindly assigned to the intervention or control group and were blind to the level of production pressure they were exposed to. They were also blinded to the purpose of the study until completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Production pressured environment (Experimental): Participants in this group were exposed to 4 audio recordings applying standardized pressure. Unlimited time.
  Interventions: Other: Production pressure
- Regular environment (No Intervention): The control group was asked to complete the same task also with unlimited time. They were not exposed to the audio recordings.

INTERVENTIONS:
Other: Production pressure — Participant exposed to production pressure
  Arms: Production pressured environment

SUMMARY:
This randomized, single blinded simulation based study investigates the impact that production pressure can have on the safety of patients undergoing regional anesthesia. We created a high fidelity scenario where anesthesiologists and trainees were to perform a single shot infraclavicular ultrasound guided block. Participants were randomly assigned to the intervention or control group. Participants assigned to the intervention group were exposed to various production pressure generating interventions. The goal of this study was to look at the impact of production pressure on patient safety by scoring anesthesiologists' and trainees' performance and examining the differences between the two groups.

DETAILED DESCRIPTION:
Sample size:

To our knowledge, no studies were performed to evaluate the impact of production pressure on anesthesiologists nor on how to emulate production pressure in a simulated environment. Although it is known that production pressure affects negatively healthcare workers' performance, it remains difficult to predict its impact on a scoring system such as the RAPS assessment tool. Therefore, we used a convenience sample based on the number of residents and staffs anesthesiologists who agreed to participate. Using the t value and the degrees-of-freedom of the unpaired t-test, the investigators calculated the effect size (r) to characterize the magnitude of the effect and evaluate if the sample size is enough to answer the research hypothesis. An r value of around 0.2 was considered a "weak" effect, 0.5 "medium", and 0.8 "strong". We intend to recruit between 10 to 20 participants in each group.

Scenario:

Participants were asked to obtain consent and perform a single shot infraclavicular ultrasound guided block on a 50 year old woman with mild COPD. The simulation took place in situ in a regional anesthesia block room. Upon entering the room, the anesthesiology evaluation was already completed. A CAE infraclavicular block simulator was installed on a simulated patient. A simulated anesthesiology nurse was also present to assist only. All preparation steps and safety measures had to be initiated by the participant. Participants in the intervention group were exposed to 4 standardized pre-recorded audio interventions, encouraging them to proceed faster. The choice of these interventions was based on articles and surveys detailing the common sources of production pressure for the anesthesiologist.

Data collection:

Performances were filmed in order to be reviewed by three regional anesthesia experts. Participants were then asked to fulfill a questionnaire in another room. This form included a validated task load index grid (NASA) to quantify the amount of stress experienced, demographic data and a realism score.

ELIGIBILITY:
Inclusion Criteria:

* To be a certified anesthesiologist or anesthesiology resident
* To have performed at least 10 regional anesthesia techniques including 5 infraclavicular blocks
* To consent to the study

Exclusion Criteria:

- To refuse to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
RAPS score | Through scenario completion (approximatively 25 minutes)
  Score obtained from regional anesthesia experts using the RAPS assessment tool, a validated tool to measure performance of a regional anesthesia technique (see reference)

SECONDARY OUTCOMES:
Time to complete the task | Through scenario completion (approximatively 25 minutes)
  Time between skin asepsis and needle withdrawal
Stress level experienced | Through scenario completion (approximatively 25 minutes)
  As measured by the NASA task load index, a validated tool to measure mental and physical stress experience during a task.
  The participant has to rate each 6 category on a continous scale of 21 points as shown below.
  Mental Demand From very low to very high Physical Demand From very low to very high Temporal demand From very low to very high Performance From perfect to failure (This scale in interpreted in a reverse way) Effort From very low to very high Frustration From very low to very high The next step for the participant is to do a pairwise comparison of each category by selection the most contributive.
  Results are presented with transformation of the 21 points to a 100 points scale as a rating from 0 to 100 ( Low to high task load) By using pairwise comparison, a weighted global result is also presented with a score from 0 to 100 (Low to high task load)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada